CLINICAL TRIAL: NCT07292142
Title: FMT in Triple Negative Breast Cancer Guided by ctDNA
Acronym: FRIDA
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FRIDA
Record Dates: First submitted 2025-11-19; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: The first participants recruited will be part of the Phase 1 or the trial until the investigators reach the target number of participants. The investigators will them open the recruitment of the Phase 2 Cohort 1, until the target number of participants is reached, and that the Phase 2 Cohort 2 will be open for recruitment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase I (Experimental): In preparation for Phase II of the protocol, Phase I of the study will evaluate the feasibility of stool and plasma sample collection at different time points in TNBC patients receiving standard of care NAT.
  Interventions: Other: No Intervention.
- Phase II - Cohort 1 (Experimental): Phase II aims to assess the safety and feasibility of adding FMT to the treatment regimen of patients with TNBC receiving standard of care neoadjuvant chemotherapy plus immunotherapy. As this FMT regimen has never been combined with chemo-immunotherapy in TNBC, the goal is to assess safety and feasibility first. Exploratory analyses of markers of tumor response (ctDNA and pCR rate) and gut microbiome will also be conducted before embarking on a larger study. Phase II will comprise two cohorts. Cohort 1 will be administering FMT before starting standard systemic anti-cancer therapy, in this case, NAT for early TNBC.
  Interventions: Drug: Fecal Microbiota Transplantation (FMT)
- Phase II - Cohort 2 (Experimental): Phase II aims to assess the safety and feasibility of adding FMT to the treatment regimen of patients with TNBC receiving standard of care neoadjuvant chemotherapy plus immunotherapy. As this FMT regimen has never been combined with chemo-immunotherapy in TNBC, the goal is to assess safety and feasibility first. Exploratory analyses of markers of tumor response (ctDNA and pCR rate) and gut microbiome will also be conducted before embarking on a larger study. Phase II will comprise two cohorts. In Cohort 2, patients with ctDNA+ persistence from baseline to post-cycle 1 NAT (high-risk of non-pCR) will receive "rescue" FMT therapy at mid-treatment of NAT.
  Interventions: Drug: Fecal Microbiota Transplantation (FMT)

INTERVENTIONS:
Drug: Fecal Microbiota Transplantation (FMT) — The investigators propose to test the safety and feasibility of altering the gut microbiome in the context of neoadjuvant therapy (NAT) for TNBC. This pilot study will assess the safety of FMT given with neoadjuvant chemo-immunotherapy and will determine the feasibility of conducting a future randomized clinical trial to test whether FMT improves the effectiveness of neoadjuvant chemotherapy and ICB in patients with TNBC.
  Arms: Phase II - Cohort 1; Phase II - Cohort 2
Other: No Intervention. — No FMT will be given in Phase I
  Arms: Phase I

SUMMARY:
Triple-negative breast cancer (TNBC) is an aggressive form of breast cancer, usually treated with chemotherapy and an immune checkpoint blockade (ICB) in the pre-operative or neoadjuvant phase. However, about 35% of tumors do not respond fully to this therapy, and patient prognosis is poor. Recent exciting data from our group and others suggest that the alteration of the gut microbiome via fecal microbiota transplantation (FMT) markedly affects the response to ICB in melanoma1-3. The investigators propose to test the safety and feasibility of altering the gut microbiome in the context of neoadjuvant therapy (NAT) for TNBC. This pilot study will assess the safety of FMT given with neoadjuvant chemo-immunotherapy and will determine the feasibility of conducting a future randomized clinical trial to test whether FMT improves the effectiveness of neoadjuvant chemotherapy and ICB in patients with TNBC.

This study will be divided into two phases. In Phase I (observational phase), the investigators propose to test the feasibility of collecting stool and plasma samples in TNBC patients treated with neoadjuvant therapy (NAT) without FMT treatment. In Phase II (interventional phase), patients will undergo the sample collection procedures as in Phase I, but in addition, the investigators will assess the safety and feasibility of FMT treatment in combination with NAT.

ELIGIBILITY:
Inclusion Criteria:

PHASE 1

* Patients must be 18 years old or older.
* Patients must have a confirmed diagnosis of TNBC (defined as estrogen receptor expression 0-10%, progesterone receptor expression 0-10%, and HER-2/neu negative (immunohistochemistry 0, 1+, or 2+ and fluorescent in-situ hybridization negative for HER-2 gene amplification) and are about to start neoadjuvant chemotherapy.
* Patients with ECOG performance of 0-2.
* Patients who are willing to provide serial stool and blood samples.
* Patients must be able to provide written informed consent
* Patients with available primary tumor biopsy tissue for molecular analysis

PHASE 2

* Patients must be 18 years old or older.
* Patients must have a confirmed diagnosis of TNBC (defined as estrogen receptor expression 0-10%, progesterone receptor expression 0-10%, and HER-2/neu negative (immunohistochemistry 0, 1+, or 2+ and fluorescent in-situ hybridization negative for HER-2 gene amplification) and are about to start neoadjuvant chemotherapy-immunotherapy.
* Patients with ECOG performance of 0-2.
* Patients must be able to provide written informed consent and understand the infectious risks associated with FMT administration.
* Ability to ingest capsules.
* Patients receiving systemic steroids at physiologic doses are permitted to enroll assuming steroid dose is not above the acceptable threshold (>10 mg prednisone daily or equivalent).

Exclusion Criteria:

PHASE 1

* Clinical or radiological evidence of metastatic disease.
* Known infection with HIV or hepatitis.
* Pregnant woman.

PHASE 2

* Previous anti-PD-1 treatment.
* Patient with a secondary malignancy.
* Pregnant or breastfeeding or expecting to conceive children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Current exposure to high-dose oral or intravenous corticosteroids (>10 mg of prednisone daily or equivalent). Patients who require intermittent use of bronchodilators or local steroid injections are not excluded from the study.
* Absolute neutrophil count <1.0 within 48 hours of planned FMT administration
* Has a diagnosis of immunodeficiency (for example, HIV or transplantation) or any other form of immunosuppressive therapy before trial treatment.
* Ongoing use of antibiotics or previous use of antibiotics one week before the FMT procedure.
* Probiotic supplements and food products labeled as containing probiotics must be discontinued a minimum of 24 hours before FMT administration and are not permitted during the course of neoadjuvant immunotherapy treatment.
* Presence of a chronic intestinal disease (for example, celiac, malabsorption, and colonic tumor).
* Presence of absolute contraindications to FMT administration, including toxic megacolon, severe dietary allergies (for example, shellfish, nuts, or seafood), and inflammatory bowel disease.
* Expected to require any other form of systemic or localized anti-neoplastic therapy other than those proposed by the study while on study.
* Has an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents. Patients with vitiligo, type I diabetes, or resolved childhood asthma/atopy are exceptions to this rule.
* A history of recent (<30 days) (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has serious concomitant illnesses, such as uncontrolled cardiovascular disease (congestive heart failure, uncontrolled hypertension, active evidence of cardiac ischemia, myocardial infarction, and severe cardiac arrhythmia), autoimmune diseases, severe obstructive or restrictive pulmonary diseases, active systemic infections, and inflammatory bowel disorders. This includes HIV or AIDS-related illness or active hepatitis B or C virus.
* Has an active infection requiring systemic therapy.
* Patient has received a live vaccine within 4 weeks before the first dose of treatment. Note that seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (for example, FluMist) are live attenuated vaccines and are not allowed.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of combining Fecal Microbial Transplantation (FMT) using intestinal bacteria existing in the stool of healthy donors with immunotherapy/chemotherapy in triple-negative breast cancer patients. | 20 months
  Toxicity assessments and concurrent medication review will occur at every visit throughout chemotherapy/immunotherapy treatment. Any adverse events after FMT administration will be followed until resolution or until judged stable by the investigator.
Feasibility of giving FMT is triple negative breast cancer patients treated with chemotherapy / immunotherapy prior surgery. | 7 months
  The feasibility of FMT in both cohorts will be determined based on the proportion of patients that completed each step of the study. The investigators will assess the proportion approached and declined, approached and consented, consented and withdrew before FMT, consented, screened and successfully took the FMT, and able and willing to provide post-FMT stool samples.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - London Health Sciences Center, London, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Jewish General Hospital, Montreal, Quebec